CLINICAL TRIAL: NCT01079585
Title: The Effect of 40gr Okara on Gastric Emptying
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Tel-Aviv Sourasky Medical Center (Other Government)
Collaborators: Nutrigal LTD (Unknown)
Allocation: Randomized | Model: Crossover | Masking: Single
Other Study IDs: TASMC-10-NV-014-CTIL
Record Dates: First submitted 2010-02-17; First posted 2010-03-03 (Estimated); Last update posted 2010-03-03 (Estimated); Status verified 2010-02

CONDITIONS: Healthy People

INTERVENTIONS:
Dietary Supplement: Nutrigal Okara - 100

SUMMARY:
The effect of 40gr Okara, on gastric emptying of standard meal (Muffin cake)

DETAILED DESCRIPTION:
This trail will be a single blinded, cross-over design. The study population will include 10 subjects. The patients will be randomly assigned to receive one of two Muffin cakes, with or without 40 grams Okara on three occasions (three visits). In two visits the subject will receive a Muffin cake with 40 grams Okara (but with similar caloric value), and in one visit a Muffin cake without Okara.

Postprandial gastric emptying time will be measured for each subject, by 13C Breath Test.

Okara is a natural water extracted food grade soy product, contains approximately 35% protein (mfb), and about 43% of dietary fibers.

ELIGIBILITY:
Inclusion Criteria:

* Healthy volunteers
* Age 20-65 years old
* Written Informed Consent

Exclusion Criteria:

* History of gastro-intestinal surgery
* On medication that may influence gastric emptying, or medication for weight loss
* Patient on PPI treatment, H2 Blockers or medication for weight loss
* Known allergies to soy
* Pregnancy or breast-feeding
* Smoking
* Athletes
* Metabolic syndrome or diabetes mellitus
* Family history of metabolic syndrome or diabetes mellitus
* Weight loss > 2 kg during two months before the study

Ages: 20 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2010-03; Primary Completion 2010-10 (Estimated); Study Completion 2010-12 (Estimated)

PRIMARY OUTCOMES:
To investigate the influence of 40 gram Okara on gastric emptying

CONTACTS AND LOCATIONS:
Locations (1):
- Tel Aviv Medical Center, Tel Aviv, Israel